CLINICAL TRIAL: NCT04285996
Title: IMaging Pilot Study of the αvβ6 Integrin Radiotracer [18F]-A20FMDV2 in PAtients With Solid Cancer Types
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10559QM
Record Dates: First submitted 2017-09-18; First posted 2020-02-26 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: Breast Cancer; Pancreatic Cancer; Head &Neck Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Pilot study: All registered patients will undergo a PET scan using [18F]-FBA-A20FMDV2.
  Interventions: Procedure: PET Scan

INTERVENTIONS:
Procedure: PET Scan
  Other Names: PET imaging using [18F]-FBA-A20FMDV2

SUMMARY:
A substance called integrin alpha v beta six (αvβ6) is found to be increased in some cancer cells and can play an important role in the development and spread of cancer. If the levels of integrin αvβ6 in cancer cells can be measured by carrying out PET scans, we might be able to identify and potentially treat tumours.

FBA-A20FMDV2 is a substance that binds or sticks to integrin αvβ6. It may therefore be possible to find and measure the amount of integrin αvβ6 in tumours. To do this a small amount of radioactivity will be attached to FBA-A20FMDV2 and carry out a scan called a Positron Emission Tomography (PET) scan. FBA-A20FMDV2 attached to radioactivity is known as [18F]FBA-A20FMDV2 or a radiotracer, as a very small amount of tracer dose is given to humans.

So far such scans have been carried out in healthy volunteers and in patients with a lung condition called idiopathic pulmonary fibrosis (IPF). This was to assess the safety of the radiotracer and how it is taken up in the body. However, such scans have not been performed in cancer patients. This study will help specifically investigate αvβ6 in patients with cancer and find out how [18F]FBA-A20FMDV2 is taken up in tumours. With this information, the ideal imaging method for patients with cancer can be developed.

DETAILED DESCRIPTION:
The epithelial specific integrin αvβ6 is not expressed by resting epithelia (1) but is up regulated in several cancers. It has been estimated that approximately 250,000 or 15% of new cancers (excluding non-melanoma skin cancers) that arise in the UK and USA combined will overexpress αvβ6 (2-4). αvβ6 plays a key role in tumour invasion and carcinogenesis. Strong expression of αvβ6 is associated with significant reduction in life expectancy in patients with colon, cervical, breast or non-small cell lung cancer (3-5). Recently, it has been shown in preclinical studies that antibody targeting of αvβ6 could suppress the growth of oral and breast cancer human xenografts and suppress breast cancer metastasis (6). Thus αvβ6 represents a biologically relevant target for anti-cancer therapy.

The proposal is to conduct this study in patients with solid tumours as αvβ6 is expressed exclusively by carcinomas, which are all solid tumours. As the utility of [18F]-FBA-A20FMDV2 in patients with cancer has not been evaluated a particular challenge with evaluation of this radiotracer in patients with cancer include potential metabolism and excretion of this radiotracer by the liver and kidney confounding the image quality for lower thoracic and abdominal tumours requiring optimisation of the imaging protocol. In addition, as the patients are likely to be unwell, it is imperative an imaging protocol that is patient-friendly in terms of the scan duration is developed. Additionally it would be ideal to confirm that the uptake of the radiotracer is indeed due to αvβ6 expression on the cancer cells. Therefore in this study, it is planned to evaluate the feasibility of performing such a study in patients with a variety of solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent prior to admission to this study.
2. Female or male aged ≥18 years
3. ECOG performance status of 0-2
4. Clinical diagnosis of a solid tumour measuring ≥1cm in the longest diameter as assessed by clinical imaging or by physical clinical evaluation.
5. Female patients of childbearing potential or male patients with female partners of child-bearing potential must agree to use adequate contraception as described in the protocol from the day of the scan and until 4 weeks after the scan
6. Haematologic indices (FBC, WBC, ANC, platelets count and haemoglobin) and biochemical indices (sodium, potassium, chloride, urea, creatinine, total protein, albumin, total bilirubin, ALP and AST) within local institutional limits.
7. Negative urine pregnancy test for female patients of childbearing potential prior to study entry1.
8. Availability of a formalin fixed, paraffin embedded (FFPE) tumour sample for central assessment.2

Exclusion Criteria:

1. Breast feeding female patients.
2. Previous or current exposure to animals that may harbour the foot and mouth disease virus FMDV2
3. Previous long-term (≥ 3 months) residence in a country where FMDV2 is endemic (such as certain areas of Africa, Asia and South America).
4. Subject feels unable to lie flat and still on their back for a period of up to 95 minutes in the PET/CT scanner.
5. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of the tracer, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of [18F]-FBA-A20FMDV2-PET imaging in patients with solid tumours. | at the time of the PET scan
  The uptake of the radiotracer by tumours and normal tissue

SECONDARY OUTCOMES:
Optimise PET scan time parameters | The outcome will be measured after each scan.
  Timing of radiotracer administration will be measured in tumour and normal tissue. Results will be presented by Time Activity Curves.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Principal Investigator — Queen Mary University of London; John Marshall, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom